CLINICAL TRIAL: NCT02316327
Title: Phase IV/II Open-label Study to Evaluate Prompt Response to Treatment With Cisplatin, Gemcitabine and Bevacizumab in Patients With Non-small Lung Cancer.
Brief Title: Open-label Study in Patients With Metastatic NSLC Treated With Cisplatin, Gemcitabine and Bevacizumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Dr. Noemi Reguart, MD, PhD, Oncologist, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMPACT; 2012-000459-15 (EudraCT Number)
Record Dates: First submitted 2014-12-05; First posted 2014-12-12 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine, cisplatin and bevacizumab (Experimental): Bevacizumab will be given by I.V infusion at the dose of 7.5 mg/kg on days 1 every 21 days
  Cisplatin 80 mg/m2 I.V on day 1
  Gemcitabine 1250 mg/m2 I.V on day 1 & 8
  Treatment cycles will be repeated every three weeks up to 6 cycles
  Bevacizumab monotherapy as maintenance allowed in non-progressive tumors
  Interventions: Drug: gemcitabine, cisplatin and bevacizumab

INTERVENTIONS:
Drug: gemcitabine, cisplatin and bevacizumab — Therapeutic
  Other Names: Avastin

SUMMARY:
RATIONALE: Classically the evaluation of response in lung cancer has been based in comparing pre & post treatment tumour volume by means of studying changes in the diameter of the selected target lesions by RECIST. The introduction of new targeted drugs creates the need of a different response assessment. Functional imaging techniques are able to study in vivo physiological processes of angiogenesis. Therefore, dynamic techniques may be more appropriate for assessing response to antiangiogenic drugs, whose mechanism of action is focused on tumor's vasculature normalization. Preliminary studies have demonstrated significant and very early changes in indirect vasculature parameters such as flow, blood volume and tumor perfusion with vascular-targeting agents. These techniques may be useful for selecting patients who are going to benefit from antiangiogenic therapy by an early evaluation of response by means of functional imaging method.

PURPOSE: IMPACT is an open-label, single arm phase II/IV study to evaluate the predictive value and early radiologic response or perfusion computed tomography (CT) in patients diagnosed with unresectable advanced, metastatic or recurrent non-squamous NSCLC treated with bevacizumab in combination with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES

Primary objective:

• To assess early tumour response (at day +7) in terms of blood flow as compared to Objective Response Rate (ORR) in terms of RECIST criteria (CR + PR) at day 42.

Secondary objectives:

* To assess early tumour response (at day +7) in terms of blood volume, mean transit time, enhancement peak, time to the enhancement peak and capillary tumour permeability as compared to ORR (CR + PR) at day 42.
* To assess tumour response (at day +42) in terms of blood flow, blood volume, mean transit time, enhancement peak, time to the enhancement peak and capillary tumour permeability as compared to ORR (CR + PR) at day 42.
* To assess tumour response (at day +7 and +42) in terms of blood flow, blood volume, mean transit time, enhancement peak, time to the enhancement peak and capillary tumour permeability as compared to PFS and OS
* Safety profile using NCI-CTC AE (version 4.0).
* To assess the efficacy in the subgroup of adenocarcinoma pts.

Outline:

Patients receive bevacizumab 7.5mg/kg IV, cisplatin 80mg/m2 and gemcitabine 1250 mg/m2 on days 1 and 8 up to 6 cycles of 21 days. Patients without progression may continue maintenance treatment with single-agent bevacizumab 7.5 mg/Kg on day 1 every 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Give the written informed consent to participate in the trial before carrying out any specific study procedure.
2. Histological or cytological non microcytic lung cancer (NMLC) and non squamous advanced locally or metastatic (IIIB/IV) lung cancer confirmation
3. Capability to take on the obligations with study protocol requirements.
4. Patients 18 years old.
5. ECOG functional status 0 or 1.
6. At least a measurable lung lesion with conventional TAC (i.e. ≥ 1cm) in at least one dimension its RECIST criteria (v.1.1) which has not been irradiated.
7. Appropriate bone marrow function.
8. Appropriate hepatic function.

10. International normalized ratio (INR) ≤ 1.5 and activate partial thromboplastin time (aPTT) ≤ 1.5 x UNL 7 days previous to the first study drug administration, unless patients have been used prophylactic anticoagulant treatment 11. Patients with brain metastasis which had been treated and also asymptomatic , they are eligible to participate in the study.

12. Female patients cannot be pregnant nor lactating. 13. Male fertile patients have to use a high effective method of contraception.

Exclusion Criteria:

1. Previous treatment with systemic chemotherapy for advance NMLC
2. Non microcytic- microcytic mix histology or adeno-squamous mix carcinomas with a predominant squamous component
3. Hemoptysis history ≥ grade 2 (defined as at least 2.5 ml of bright red blood) in a period of 3 months prior to receive the study drugs
4. Surgery (including open biopsy) or significant traumatic injury in a period of 28 day prior to receive the study drugs.
5. Minor surgery including a catheter insertion in a period of 24h prior to the first infusion of bevacizumab
6. Proof that the tumor can compress or invade a main vessel in image tests
7. Radiotherapy in any site for any reason in a period of 28 days prior to receive the study drugs. It is permitted palliative radiotherapy to bone lesions .
8. Aspirin based medication (> 325 mg/day or clopidogrel > 75mg/day) present or recent (in a period of 10 days from the first bevacizumab infusion). Medication with oral anticoagulants agents or parenteral medication on full doses (e.g. in a therapeutic range) or the use of thrombolytic agents with present and recent therapeutic intentions (in a period of 10 days prior to the first bevacizumab infusion). The prophylactic medication with anticoagulants is permitted
9. History or evidence of inheritance bleeding diathesis or coagulopathy with bleeding risk
10. Active gastrointestinal bleeding
11. Inadequate controlled hypertension .
12. Cardiovascular disease .
13. Wounds that do not heal, active peptide ulcer or non treated bone fractures.
14. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess in the 6 months prior to receive the study drugs
15. Known hypersensitivity to bevacizumab, cisplatin or gemcitabine or any of its excipients
16. Important known hypersensitivity to iodated contrast agents
17. Another neoplastic disease other than NMLC in a period of 5 years prior to receive the study drugs with exemption of in situ cervix carcinoma, basal or squamous skin cancer, prostate cancer treated with curative intention and in situ breast ductal carcinoma treated with curative intention
18. Proof of any other disease, neurologic or metabolic dysfunction, lab abnormality or physical test that can reasonably make suspect circumstances that would contraindicate the use of a certain investigational or the standard treatment used in this study or that puts the patient into a greater risk to suffer complications related to the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-07; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
To evaluate blood supply, blood volume, time to peak flow increase and permeability and relation with the objective response to treatment (RC+RP) | The results on baseline and day 7 to treatment in terms of blood suply, blood volume, time of peak flow increase and permeability and relation with the objective (RC+RP) at day 42.

SECONDARY OUTCOMES:
To evaluate the response to treatment in terms of blood supply, blood volume and time to peak flow increase and permeability. | To evaluate at day +42 the response to treatment in terms of blood supply, blood volume and time to peak flow increase and permeability.
To evaluate the blood supply, blood volume, time to peak flow increase, permeability related with PFS and OS. | To evaluate the blood fluid, blood volume, time to peak flow increase, permeability at baseline visita related with PFS and OS.
To evaluate the response to treatment at day +7 and +42 in terms of blood fluid, blood volume, time to peak flow increase, permeability at baseline visit related with PFS and OS. | To evaluate the response to treatment at day +7 and +42 in terms the blood fluid, blood volume, time to peak flow increase, permeability at baseline visita related with PFS and OS.
The safety of the treatment following NCI-CTC AE (version 4.0) | The safety of the treatment following NCI-CTC AE (version 4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Noemi Reguart, MD, PhD, Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Background] Reck M, von Pawel J, Zatloukal P, Ramlau R, Gorbounova V, Hirsh V, Leighl N, Mezger J, Archer V, Moore N, Manegold C. Phase III trial of cisplatin plus gemcitabine with either placebo or bevacizumab as first-line therapy for nonsquamous non-small-cell lung cancer: AVAil. J Clin Oncol. 2009 Mar 10;27(8):1227-34. doi: 10.1200/JCO.2007.14.5466. Epub 2009 Feb 2. PMID 19188680
- [Background] Tacelli N, Remy-Jardin M, Copin MC, Scherpereel A, Mensier E, Jaillard S, Lafitte JJ, Klotz E, Duhamel A, Remy J. Assessment of non-small cell lung cancer perfusion: pathologic-CT correlation in 15 patients. Radiology. 2010 Dec;257(3):863-71. doi: 10.1148/radiol.10100181. Epub 2010 Sep 15. PMID 20843993
- [Background] Fraioli F, Vetere S, Anile M, Venuta F. Computed tomography perfusion: a new method to evaluate response to therapy in lung cancer. J Thorac Oncol. 2011 Sep;6(9):1599-600. doi: 10.1097/JTO.0b013e3182259207. No abstract available. PMID 21849856
- [Background] Tacelli N, Santangelo T, Scherpereel A, Duhamel A, Deken V, Klotz E, Cortot A, Lafitte JJ, Wallyn F, Remy J, Remy-Jardin M. Perfusion CT allows prediction of therapy response in non-small cell lung cancer treated with conventional and anti-angiogenic chemotherapy. Eur Radiol. 2013 Aug;23(8):2127-36. doi: 10.1007/s00330-013-2821-2. Epub 2013 Apr 4. PMID 23553586
- [Background] Yuan X, Zhang J, Quan C, Cao J, Ao G, Tian Y, Li H. Differentiation of malignant and benign pulmonary nodules with first-pass dual-input perfusion CT. Eur Radiol. 2013 Sep;23(9):2469-74. doi: 10.1007/s00330-013-2842-x. Epub 2013 Jun 22. PMID 23793548